CLINICAL TRIAL: NCT07070024
Title: Efficacy of Microneedling With Vitamin C in Performing Gingival Depigmentation Compared With Conventional Scalpel and Diode Laser: A Randomized Controlled Trial
Brief Title: Efficacy of Microneedling With Vitamin C in Performing Gingival Depigmentation
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Asmaa Eid Ragab Abdelal, Resident at oral medicine and periodontology department Fayoum university, Fayoum University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: gingival depigmentation
Record Dates: First submitted 2025-05-13; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Gingival Pigmentation
MeSH Terms: interventions — Ascorbic Acid; Percutaneous Collagen Induction; Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: MN will be achieved using a Dermapen device. *** c) The device allows for adjustable penetration depth, ranging from 0.2 mm to 3 mm, based on the gingival thickness. d) The needle tip comprises 12 to 24 needles arranged in rows, providing six-speed modes that span from 412 cycles/min at the lowest speed to 700 cycles/min at the highest speed. e) The Dermapen will be positioned perpendicular to the gingival surface, and microneedling will be executed horizontally, vertically, and diagonally approximately four to five times f) Across the entire hyperpigmented gingival surface until subtle microbleeding and mild erythema became evident. g) Topical ascorbic acid powder ****, (1,000 mg/mL) mixed with saline will be applied over the gingiva for 10 minutes. h) Each individual will be undergoing a total of three treatment sessions of microneedling, spaced out by 10 days
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Microneedling with vitamin C (Active Comparator): Prior to the MN procedure, local infiltration anesthesia will be administered as used in control group b) MN will be achieved using a Dermapen device. *** c) The device allows for adjustable penetration depth, ranging from 0.2 mm to 3 mm, based on the gingival thickness. d) The needle tip comprises 12 to 24 needles arranged in rows, providing six-speed modes that span from 412 cycles/min at the lowest speed to 700 cycles/min at the highest speed. e) The Dermapen will be positioned perpendicular to the gingival surface, and microneedling will be executed horizontally, vertically, and diagonally approximately four to five times f) Across the entire hyperpigmented gingival surface until subtle microbleeding and mild erythema became evident. g) Topical ascorbic acid powder ****, (1,000 mg/mL) mixed with saline will be applied over the gingiva for 10 minutes. h) Each individual will be undergoing a total of three treatment sessions of microneedling, spaced out by 10 days
  Interventions: Drug: Vitamin C; Device: Microneedling
- Diode laser (Active Comparator): Topical anesthetic spray will be applied to the operating area. Energy output, pulse duration, and focal distance will be determined based on manufactures instruction. b) Patient, doctor and assistant will wear protective glass before starting the procedure. c) Depigmentation will be carried out using semiconductor Sirolaser BlueWith proper isolation, depigmentation procedure will be done. e) Laser ablation will be started from the mucogingival junction toward the free gingival margin, including interdental papilla. f) The laser beam will be applied using the "brush technique," as described by Tal (Tal et al.,2003) and the tip will be kept in motion all the time. g) Remnants of the ablated tissue will be removed using sterile gauze dampened with saline solution
  Interventions: Device: Diode laser
- scalpal surgery (Active Comparator): Local anesthesia will be administered through infiltration (2% lidocaine with epinephrine 1:100,000) * at the surgical site. b) Employing surgical blade number 15c, the gingival epithelium in the pigmented area will be excised. c) The blade will be oriented roughly parallel to the elongated axis of the teeth. d) A meticulous assessment of the revealed connective tissue surface will be performed, and any residual tissue tags will be removed with surgical scissors. e) Hemorrhage control will be managed by applying a pressure pack, and after achieving hemostasis, a periodontal dressing (a non-eugenol zinc oxide dressing) will be administered to cover the wound for one week
  Interventions: Procedure: scalpal

INTERVENTIONS:
Drug: Vitamin C — Topical ascorbic acid powder, (1,000 mg/mL) mixed with saline will be applied over the gingiva for 10 minutes.
  Arms: Microneedling with vitamin C
Device: Microneedling — MN will be achieved using a Dermapen device. c) The device allows for adjustable penetration depth, ranging from 0.2 mm to 3 mm, based on the gingival thickness. d) The needle tip comprises 12 to 24 needles arranged in rows, providing six-speed modes that span from 412 cycles/min at the lowest speed to 700 cycles/min at the highest speed. e) The Dermapen will be positioned perpendicular to the gingival surface, and microneedling will be executed horizontally, vertically, and diagonally approximately four to five times f) Across the entire hyperpigmented gingival surface until subtle microbleeding and mild erythema became evident Each individual will be undergoing a total of three treatment sessions of microneedling, spaced out by 10 days
  Arms: Microneedling with vitamin C
Device: Diode laser — Energy output, pulse duration, and focal distance will be determined based on manufactures instruction. b) Patient, doctor and assistant will wear protective glass before starting the procedure. c) Depigmentation will be carried out using semiconductor Sirolaser Blue With proper isolation, depigmentation procedure will be done. e) Laser ablation will be started from the mucogingival junction toward the free gingival margin, including interdental papilla. f) The laser beam will be applied using the "brush technique," as described by Tal (Tal et al.,2003) and the tip will be kept in motion all the time. g) Remnants of the ablated tissue will be removed using sterile gauze dampened with saline solution
  Arms: Diode laser
Procedure: scalpal — Employing surgical blade number 15c, the gingival epithelium in the pigmented area will be excised. c) The blade will be oriented roughly parallel to the elongated axis of the teeth. d) A meticulous assessment of the revealed connective tissue surface will be performed, and any residual tissue tags will be removed with surgical scissors. e) Hemorrhage control will be managed by applying a pressure pack, and after achieving hemostasis, a periodontal dressing (a non-eugenol zinc oxide dressing) will be administered to cover the wound for one week.
  Arms: scalpal surgery

SUMMARY:
The present study will be carried to clinically evaluate the efficacy of microneedling with vitamin C in performing gingival depigmentation in comparison with conventional scalpel and diode laser.

DETAILED DESCRIPTION:
Gingival depigmentation can be considered a periodontal plastic procedure, whereby the gingival hyperpigmentation is removed by various techniques where the technique selection should primarily be based on clinical experiences and individual preferences with primary indication of demand for improved esthetics. Different techniques for depigmentation include: Scalpel technique, Cryosurgery, Electrosurgery, Lasers as neodymium-doped yttrium aluminum garnet (Nd: YAG), Erbium-doped yttrium-aluminum-garnet (Er: YAG) laser, Carbon dioxide laser CO2 and diode laser. also, Chemical methods including acoustic agents (not used nowadays) was used for treatment of gingival pigmentation. Other methods as free gingival graft and acellular dermal matrix allograft can also be used where the aim is masking the pigmented gingiva. Diode laser is a high-power semiconductor laser that emits energy at a wavelength between 800 and 1000 nm. It has an affinity for hemoglobin and melanin; therefore, it is more efficient and better equipped to address deeper soft tissue problems. It is indicated for cutting and coagulatinggingiva and oral mucosa, creating zones of thermal necrosis of less than 1 mm and hemostasis of the affected mucosa. It has been reported as effective, pleasant and reliable method with minimal postoperative discomfort, less bleeding, low recurrent rate and faster wound healing for depigmentation procedure. The light of this laser is emitted through synthetic sapphire tips in contact mode then transmitted to optical fibers to etch or vaporize soft tissues. Vitamin C , also known as ascorbic acid, is a water-soluble vitamin that has significant antioxidant properties that protects cells from free radical damage. In addition, vitamin C also nurtures the growth and repair of skin, cartilage, bone, and teeth. Vitamin C was reported to be effective in reducing melanogenesis directly and thus promoting depigmentation. This is accomplished by interacting with tyrosinase, leading to the suppression of tyrosinase enzyme activity and, consequently, a reduction in melanin production. Vitamin C affects melanocyte function rather than the number, when compared with other approaches that relying on the destruction of melanocytes. The food and drug administration (FDA) has legally authorized microneedling (MN) devices to improve the appearance of facial acne scars, facial wrinkles, and abdominal scars. However, there are various types of MN devices including dermaroller, dermastamp, and dermapen. Dermapen is the only device that can be applied intraorally due to its small size and changeable head. This increases the accessibility inside the mouth and makes it easy to be used for a larger number of patients. This device is a wireless electric device with automated features that allow the operator to modify the speeds, pressures, and depth of penetration. It was necessary to generate precise bleeding pinpoints by MN to achieve optimal results. These microholes allow the therapeutic medication to penetrate easily into the connective tissues, stimulating new collagen production and affecting melanocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with bilateral, diffuse and symmetric physiologic gingival pigmentation in the labial maxillary or mandible gingiva.
2. Patients free from any systemic diseases according to criteria of Modified Cornell Medical Index. (Abramson J et al., 1966)
3. Periodontally healthy patient.
4. Patients with age between 18 and 50 years

Exclusion Criteria:

1. Smokers.
2. Drugs intake "mainly those associated with gingival pigmentation".
3. Pregnant and lactating women.
4. Patients with thin gingival phenotype "with scalpel group".
5. Gingival pigmentation associated with occupational hazards.
6. Individuals undergoing chemotherapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the efficacy of gingival depigmentation. | baseline , 3 months , 6 months
  The primary outcome is the assessment of how well the treatment removes or reduces the appearance of dark (pigmented) areas on the gums. This is often evaluated using a standardized index like the Degree of Oral Pigmentation Index (DOPI).
  The efficacy of different techniques ( surgical scalpal, laser, microneedling with vitamin C is then compared based on the degree of pigmentation reduction achieved and the rate of repigmentation over time Degree of gingival pigmentation will be done using Oral Pigmentation
  Index (Dummett et al ;1964) as following:
  (0) pink tissue, no clinical pigmentation.
  1. mild light brown tissue, mild clinical pigmentation.
  2. medium brown or mixed brown and pink tissue, moderate clinical pigmentation.
  3. deep brown/blue-black tissue, heavy clinical pigmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Ahmed Dr/ Rehab Ahmed Osman, Lecturer, Study Director — faculty of dentistry Fayoum university

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] P SM, S S. Comparative Assessment of Gingival Depigmentation Using Scalpel Versus Microneedling With Ascorbic Acid: A Randomized Controlled Trial. Cureus. 2024 Apr 15;16(4):e58285. doi: 10.7759/cureus.58285. eCollection 2024 Apr. PMID 38752063
- [Background] Murthy MB, Kaur J, Das R. Treatment of gingival hyperpigmentation with rotary abrasive, scalpel, and laser techniques: A case series. J Indian Soc Periodontol. 2012 Oct;16(4):614-9. doi: 10.4103/0972-124X.106933. PMID 23493062
- [Background] Mostafa D Sr, A Alaizari N, M AlOtaibi S, Ahmed Aldosari N, Rabie Al-Anazi J, S Alsughayer R, M AlFayir H, S AlHarthi M, H AlAnazi M. Gingival Depigmentation Using Microneedling Technique With Topical Vitamin C: A Prospective Case Series. Cureus. 2023 Feb 23;15(2):e35345. doi: 10.7759/cureus.35345. eCollection 2023 Feb. PMID 36974245
- [Background] Abramson JH. The cornell medical index as an epidemiological tool. Am J Public Health Nations Health. 1966 Feb;56(2):287-98. doi: 10.2105/ajph.56.2.287. No abstract available. PMID 5948222